CLINICAL TRIAL: NCT03301025
Title: Pregabalin Effects on Hypotensive Anesthesia During Spine Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa Mazy Mazy, Associate professor of anesthesia and surgical intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R/17.07.107
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Spine Surgery
Keywords: Pregabalin, hypotensive anesthesia, blood loss, analgesia
MeSH Terms: conditions — Hemorrhage; Agnosia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin group (Active Comparator): (n=53):
  Interventions: Drug: Pregabalin
- placebo group (Placebo Comparator): (n=53):
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150 mg capsule, one h preinduction of general anesthesia
  Other Names: (LYRICA® 150 mg capsule- PFIZER)
  Arms: Pregabalin group
Drug: placebo — given a placebo identical capsule once one hour before anesthesia
  Other Names: control
  Arms: placebo group

SUMMARY:
Elective lumbar spine surgical procedures are commonly performed under controlled hypotension during general anesthesia. That is beneficial to limit the intraoperative blood loss and transfusions and improves surgical field. Deliberate hypotension could be achieved via various medications but mostly associated with significant side effects. Pregabalin effectively augmented hypotensive anesthesia. The hypothesis is that Pregabalin 150 mg single preoperative dose may augment intraoperative deliberate hypotension that will be reflected on blood loss and nitroglycerin consumption.

DETAILED DESCRIPTION:
An arterial line will be established then general anesthesia will be conducted. After adequate preoxygenation, anesthesia induction by IV fentanyl 1.5µg/kg, propofol 2 mg/kg, and atracurium 0.5 mg/kg then appropriated size tracheal tube. The ventilator settings will be adjusted to maintain the end-tidal carbon dioxide tension (ETco2) at 30-35 mm Hg. Anesthesia will be maintained by isoflurane concentration 1.2%, with 40% oxygen in air then IV infusion of fentanyl 0.05 mcg/kg/min was started while atracurium 0.1 mg/kg incremental dose as required. Then patients will be turned into the prone position above pad support permitting free hanging of the abdomen. Intraoperatively, the target mean arterial arterial blood pressure (MBP) is 55-65 mm Hg. After surgical incision, if MBP exceeds 65 mm Hg (defined as hypertension) it will be managed by: increasing isoflurane MAC up to 2%, if no response after 5 min, Nitroglycerin infusion initiated at 0.5 mcg/kg/min to 40 mcg/kg/min. Hypotension (MBP <55 mm Hg) will be treated by stopping nitroglycerin, proper compensation of losses, reducing Isoflurane MAC. If persisted; vasoactive drugs will be used. Bradycardia (HR <50 beat/min.), treated with 0.01 mg/kg atropine IV increments.

The nitroglycerin infusion will be stopped after the finial surgical hemostasis. Fentanyl infusion will be stopped before ligament sutures. Isoflurane will be closed after the last surgical suture. After dressing, patient will be turned to the supine position and morphine 0.025 mg/kg IV will be administered then 0.04 mg/kg neostigmine and 0.015 mg/kg atropine for reversal. Extubation will be done after establishment of acceptable spontaneous respiration.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score I-II
* admitted to undergo lumbar discectomy or spinal fixation surgery under general anesthesia

Exclusion Criteria:

* Patients on anti-hypertensive treatment, diuretics, corticosteroids, pregabalin, gabapentin, anticonvulsants, antipsychotics,
* alcohol addiction or drug abuse
* patients with history of allergy to any drug used in the study .
* pregnant or nursing women
* patients with peripheral neuropathy, endocrinal diseases, bleeding abnormality,
* cardiac, hepatic or renal impairment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Nitroglycerin consumption | Intraoperative
  the total nitroglycerin consumption in milligram to maintain the target mean arterial pressure (MAP) 55- 65 mmHg.

SECONDARY OUTCOMES:
Estimated blood loss | intraoperative
  towels are weighted, plus suction volume without irrigation fluids in milliter.
The number of transfused blood unites | intraoperative
  Packed red blood cell unites
heart rate (HR) | Basal, during intubation, then at 1, 5, 30, 60, 90, 120, 150, 180, 210 minutes post extubation, then postoperatively at 1 and 2 hours.
  in beat/min
end-tidal isoflurane concentration | at 30, 60, 90, 120, 150 , 180, 210 minutes after intubation.
  in percent
Surgeon satisfaction about the field | within 2 hours from the end of surgery.
  using a six-point scale (0 = no bleeding, virtually bloodless field; 5 = uncontrolled) bleeding).
Sedation | at 0, 2, 4, 6, 12, 24 hours postoperatively
  (Ramsay sedation scale)
The time to the first request of analgesia. | 24 hours postoperative
  in hours
Postoperative pain | at 0, 2, 4, 6, 12, 24 hours postoperatively.
  (VAS 0-10 scale) 10 is the worst pain
The total morphine consumption | in the 1st 24 hours postoperatively
  in mg
Frequency of adverse effects | during the first 24 hours postoperatively
  dizziness, headache, nausea and vomiting, or pruritus.
Peak airway pressures | 10 minutes after settled prone position
  in centimeter water
invasive mean arterial blood pressure (MAP) | Basal, during intubation, then at 1, 5, 30, 60, 90, 120, 150, 180, 210 minutes post extubation, then postoperatively at 1 and 2 hours.
  in millimeter mercury (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Mazy, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (2):
- Egypt (2):
  - Delta Hospital, Al Mansurah, Dakahlia Governorate
  - Mansoura University Hospital, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Yes
all data will be available after about 6 months
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: e mail: alaa_mazy@yahoo.com
URL: http://alaa_mazy@yahoo.com